CLINICAL TRIAL: NCT03935477
Title: An Observational Study of Tissue Oxygen Monitoring for Detecting Impending Shock States in the Critically Ill and Those Undergoing High Risk Surgery
Brief Title: Surrogate of Adequate Perfusion: Bladder Tissue Oxygen Monitoring
Acronym: SoAP-BOx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: Wellcome Trust (Other); Department of Health, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Professor Mervyn Singer, Clinical Professor, University College London Hospitals
Other Study IDs: CIP_DPW016_OBS
Record Dates: First submitted 2019-03-13; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-05

CONDITIONS: Shock; Sepsis; Surgery
MeSH Terms: conditions — Shock; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk surgery: those undergoing elective and emergency, high-risk surgery receiving arterial cannulation and urethral catheterisation as standard
  Interventions: Device: WellBeing catheter
- Critical Care: Emergency admissions to UCLH critical care unit receiving arterial cannulation and urethral catheterisation as standard
  Interventions: Device: WellBeing catheter

INTERVENTIONS:
Device: WellBeing catheter — Urethral catheterisation with integral Wellbeing Catheter to measure bladder tissue oxygen tension

SUMMARY:
The extent and duration of tissue hypoxia is a major determinant of outcome following major, high-risk surgery and in critical illness. Prompt restoration of tissue oxygenation through resuscitation in all likelihood improves outcomes. There are currently no bedside monitors in clinical practice that track tissue perfusion per se, instead clinicians rely on crude surrogates such as heart rate and blood pressure, urine output, serum lactate of global flow (cardiac output) monitoring.

This is a first-in-man trial of a new device to measure tissue oxygenation in real time in a major, high-risk surgical and critical care cohort. The device consists of an oxygen sensing probe incorporated into a modified urinary catheter, which relies on photoluminescence technology and the quenching properties of oxygen.

Once inserted, the drained bladder collapses round and envelopes the probe which continuously measures tissue oxygenation of the bladder urothelium.

The investigators hope to (i) Establish that tissue oxygenation can be safely monitored using this technology, deployed in this way. (ii) Define a normal range for bladder tissue oxygenation in man as measured using this device. (iii) Compare tissue oxygenation against other markers of perfusion status in current clinical practice and assess its performance at detecting inadequate perfusion against these other modalities. (iv) assess the diagnostic and prognostic capabilities of the tissue oxygenation monitoring at detecting hypo-perfusion and predicting outcome. (v) Further assess the tissue response to an 'oxygen challenge' in identifying occult hypo-perfusion. (vi). Provide pilot work required to inform future, interventional studies where similar patients would be resuscitated to tissue oxygenation targets alongside routine clinical practice.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* having major elective or emergency surgery (deemed to need invasive BP monitoring by anaesthetist) and a urinary catheter
* OR emergency admission to critical care (necessitating arterial line and urinary catheter).

Exclusion Criteria:

* age <18
* pregnancy
* contraindication to arterial cannulation or urethral catheterisation
* surgery on lower urinary tract/bladder
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: as described above
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Time to identification of a low bladder tissue PO2 versus time to development of hyperlactatemia (2 mmol/l) | Up to 7 days
  Comparison of bladder tissue PO2 values (normal range to be defined as part of this first-in-man study) against lactate values >2 mmol/l
Time to identification of a low bladder tissue PO2 versus time to development of hypotension (mean BP <60 mmHg) | Up to 7 days
  Comparison of bladder tissue PO2 values (normal range to be defined as part of this first-in-man study) against mean BP values <60 mmHg

SECONDARY OUTCOMES:
Number of Participants With Device-Related Adverse Events | Up to 28 days
  Monitoring of direct device-related complications (e.g. bleeding, bladder perforation)
Identification of future complications in postoperative patients | Up to 7 days
  Low bladder tissue PO2 values identify postoperative complications using POMS-score-defined morbidity at Days 3 and 7

CONTACTS AND LOCATIONS:
Overall Officials: Mervyn Singer, MD, Principal Investigator — UCL
Locations (1):
- UCL Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No